CLINICAL TRIAL: NCT06432465
Title: tDCS to Decrease Opioid Relapse (UH3)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1317333; 4UH3DA047793 (NIH)
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Opioid Use Disorder
Keywords: opioid craving; buprenorphine; methadone; EEG; transcranial direct current stimulation
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- active tDCS (Active Comparator): Each participant will undergo 5 consecutive (i.e., business days) sessions of active tDCS delivered to the DLPFC. During each session, participants are engaging in tasks that activate the cognitive control network.
  Interventions: Device: active tDCS
- sham tDCS (Sham Comparator): Each participant will undergo 5 consecutive (i.e., business days) sessions of sham tDCS delivered to the DLPFC. During each session, participants are engaging in tasks that activate the cognitive control network.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — The anode will be placed over the right DLPFC (F4 on the EEG 10-20 system) and the cathode over the left DLPFC65 (F3) using 25cm2 sponges at an intensity of 2mA. Stimulation will be delivered for 20 minutes via two saline-soaked surface sponge electrodes and a battery-driven, constant current stimulator (NeuroConn DC Stimulator Plus).
  Arms: active tDCS
Device: sham tDCS — Same device and procedures as active tDCS with the exception that the device includes a study mode, in which subject-specific codes are entered to deliver active or sham stimulation, keeping the administrator blinded. Sham stimulation will use a method in which stimulation will be ramped up and back down over a 30-second period at the beginning and end of sham tDCS.
  Arms: sham tDCS

SUMMARY:
Investigators will measure behavioral and brain responses following transcranial direct current stimulation (tDCS) to the dorsolateral prefrontal cortex (DLPFC) (anode on right DLPFC, cathode on the left DLPFC) delivered during cognitive control network (CCN) priming. In Phase I, the EEG provided validation of expected changes in these networks following tDCS stimulation of the DLPFC. In this current phase (II), the investigators will perform a larger randomized clinical trial (RCT) (active vs. sham control) to address long-term neurobehavioral outcomes, including opioid relapse, craving, and sustained EEG changes.

DETAILED DESCRIPTION:
Investigators will perform an RCT in 100 opioid dependent participants who recently initiated buprenorphine or methadone. Participants will be randomized to receive five sessions of tDCS+CCN priming stimulation vs. sham tDCS+CCN priming. Participants will be assessed three times using electroencephalographic (EEG), once prior to tDCS+CCN priming, right after the completion of 5 sessions of tDCS+CCN priming (one week later), and again 10 weeks later.

This phase will address long-term (3- and 6-month) neurobehavioral outcomes, including opioid relapse, craving, and sustained EEG changes during a paradigm that challenges networks associated with craving (CR) and cognitive control (CCN). During the 24 weeks of buprenorphine or methadone maintenance treatment, the investigators will examine our primary clinical outcome, relapse (opioid use on >4 days per month and having an opioid positive urine screen), as well as days of opioid use.

ELIGIBILITY:
Inclusion Criteria:

1. current opioid dependence
2. between 21-60 years of age
3. recent initiation of buprenorphine or methadone (≤30days)
4. enrolled in Butler Hospital's Alcohol and Drug Inpatient Unit, Alcohol and Drug Partial Hospital Treatment Program, Intensive Outpatient Services, or Outpatient Services at Butler Hospital OR receive opioid-treatment services in the community.

Exclusion Criteria:

1. current diagnosis of organic brain disorder (e.g., Parkinson's disease, Huntington's disease, multiple sclerosis, intracranial mass/infection, hydrocephalus)
2. bipolar, schizophrenia, schizoaffective, or schizophreniform disorder, or current psychosis associated with any disorder
3. current suicidality
4. evidence of significant neurocognitive dysfunction
5. conditions associated with heightened tDCS risks, e.g., seizure disorder, nonremovable intracranial metal objects (other than dental fillings and dental implants), skin disease or active lesions on the scalp, migraine/other headache disorder with significant active symptoms, traumatic brain injury or skull fracture within the past year, any implanted medical devices or device components that can interact with electromagnetic fields or are controlled by physiological signals
6. probation/parole requirements or an upcoming move that might interfere with protocol participation
7. planning to terminate buprenorphine or methadone in less than 3 months
8. current pregnancy or plan to become pregnant in the next month.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid Craving | 2 weeks
  Modified Penn Alcohol Craving (0 = no craving to 30 = extreme craving)

SECONDARY OUTCOMES:
EEG theta activity | 2 weeks
  theta event rate during working memory task
opioid relapse | 24 weeks
  Timeline Follow back

CONTACTS AND LOCATIONS:
Overall Officials: Abrantes Abrantes, Ph.D., Principal Investigator — Butler Hospital; Michael Stein, M.D., Principal Investigator — Boston University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared online at ICPSR.
Time Frame: 1-year after the end of the study